CLINICAL TRIAL: NCT02720965
Title: Effect of Perineural Catheter Analgesia on Patient Experience After Orthopedic Surgery
Brief Title: Remote Controlled Analgesia on Patient Experience
Acronym: R-CAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9677
Record Dates: First submitted 2016-03-22; First posted 2016-03-28 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2016-03

CONDITIONS: Orthopaedic Surgery
Keywords: Pain Acute; Orthopedic Surgery; Satisfaction Nerve Blocks
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Electronic pump (Experimental): Continuous nerve blocks Remote-controlled perineural local anesthetics delivery
  Interventions: Other: Remote-controlled perineural local anesthetics delivery
- single injection (No Intervention): single injection

INTERVENTIONS:
Other: Remote-controlled perineural local anesthetics delivery — Remote-controlled perineural local anesthetics delivery
  Arms: Electronic pump

SUMMARY:
The main objective of this study is to compare the efficacy of continuous nerve blocks with single injection in terms of perioperative patient satisfaction after scheduled orthopedic ambulatory surgery. Subgroup analyses will be performed, a priori, according to patients Pain Catastrophizing Scale (PCS) and type of surgery.

Secondary objectives comprise the assessment of pain, readmission rates, patient mobilization, quality of sleep and heart rate collected by an activity tracker. Scales about quality of recovery will be performed on day 1, about quality of life on day 45 and presence of neuropathic pain will be screened at 3 months. An economic study will also be conducted, including work resumption at 3 months.

This is a multicentric prospective study. Three hundred patients will be randomized in two parallel groups: continuous nerve blocks delivered thru remote-controlled electronic pump versus single local anesthetics injection.

The primary endpoint is the EVAN-G patient satisfaction scale, scored at day 2. Secondary endpoints will include assessment of pain, opiates consumption, sensitivity and motricity scores, rate of catheter falls at home, hospital readmission, patient mobilization, sleep and heart rate as assessed by an activity tracker, PCS before the surgery and Quality of Recovery (QoR-40) scale at day 1, Short-Form 36 (SF36) at day 45 and Neuropathic Pain assessment (DN4) at day 90.

DETAILED DESCRIPTION:
Acute postoperative pain is poorly treated. More than three-quarters of patients complain of pain, from moderate to extreme, after surgery. In orthopedic surgery, continuous nerve blocks analgesia has proved effective among in-hospital patients but single injection strategy is easier to implement in the growing outpatient setting.

The main objective of this study is to compare the efficacy of continuous nerve blocks with single injection in terms of perioperative patient satisfaction after scheduled orthopedic ambulatory surgery. Subgroup analyses will be performed, a priori, according to patients Pain Catastrophizing Scale (PCS) and type of surgery.

Secondary objectives comprise the assessment of pain, readmission rates, patient mobilization, quality of sleep and heart rate collected by an activity tracker. Scales about quality of recovery will be performed on day 1, about quality of life on day 45 and presence of neuropathic pain will be screened at 3 months. An economic study will also be conducted, including work resumption at 3 months.

The inclusion criteria are adults undergoing outpatient scheduled orthopedic surgery under general anesthesia with regional analgesia.

Non-inclusion criteria are patients over 80 years, documented cognitive impairment, inability to complete a self-administered questionnaire, presenting American Society of Anesthesiology (ASA) physical status 3 unsteady or 4, or spontaneously requiring analgesic perineural catheter or a single injection of local anesthetics.

This is a multicentric prospective study. Three hundred patients will be randomized in two parallel groups: continuous nerve blocks delivered thru remote-controlled electronic pump versus single local anesthetics injection.

The primary endpoint is the EVAN-G patient satisfaction scale, scored at day 2. Secondary endpoints will include assessment of pain, opiates consumption, sensitivity and motricity scores, rate of catheter falls at home, hospital readmission, patient mobilization, sleep and heart rate as assessed by an activity tracker, PCS before the surgery and Quality of Recovery (QoR-40) scale at day 1, Short-Form 36 (SF36) at day 45 and Neuropathic Pain assessment (DN4) at day 90.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject aged 18 or more, up to 80 years;
* Undergoing potentially painful scheduled orthopedic surgery under general anesthesia.
* Eligible to outpatient care;
* Respecting the ambivalence clause defined below:

  1. no cons-indication to analgesic perineural catheter;
  2. not known allergy to local anesthetics;
  3. likely to be a candidate for continuous nerve block analgesia;
* Ability to complete a self-reported questionnaire;
* Have given written informed consent

Exclusion Criteria:

* Age less than 18 or more than 80 years;
* Pregnant or nursing women ;
* Not being affiliated to the social security scheme;
* Known allergy to local anesthetics of the amide type;
* Regulatory constraints in the outpatient management of perineural catheters not respected:

  1. Inability of daily nursing care;
  2. No presence of a responsible adult at home the night of the intervention;
* Scheduled hospital stay;
* ASA physical status score (American Society of Anesthesiologists) above 3 or 3 unsteady;
* Spontaneous request for continuous nerve block or single injection;
* Topic unable to fulfill only a self-administered questionnaire (inability to read French, severe cognitive impairment);
* Subject with cognitive impairment already documented (Alzheimer, dementia, neurological sequelae);
* Topic treated with antipsychotics (neuroleptics or lithium);
* Subject has a documented chronic pain syndrome;
* Active consumer of narcotic topic;
* Topic have not signed informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2016-06-07 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2019-12-02 (Actual)

PRIMARY OUTCOMES:
Patient experience and satisfaction scale (EVAN-G) | Second day after surgery
  Description: Patient experience and satisfaction scale

SECONDARY OUTCOMES:
Patient quality of recovery (QoR) | First day after surgery
  Description: Patient quality of recovery

CONTACTS AND LOCATIONS:
Overall Officials: Xavier CAPDEVILA, M.D., Ph.D., Study Chair — University Hospital, Montpellier
Locations (1):
- Department of Anesthesiology and critical care, Lapeyronie University Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Maurice-Szamburski A, Grillo P, Cuvillon P, Gazeau T, Delaunay L, Auquier P, Bringuier S, Capdevila X. Comparison of continuous with single-injection regional analgesia on patient experience after ambulatory orthopaedic surgery: a randomised multicentre trial. Br J Anaesth. 2022 Sep;129(3):435-444. doi: 10.1016/j.bja.2022.05.039. Epub 2022 Jul 7. PMID 35811140